CLINICAL TRIAL: NCT01723631
Title: Study Multicenter, Controlled, Prospective, Non-randomized Test to Analyze the Myelin-TRAP as Diagnostic Tool in Multiple Sclerosis
Brief Title: Analyze the Myelin-TRAP as Diagnostic Tool in Multiple Sclerosis
Acronym: TRAP-Myéline
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The number of patients achieved is sufficient to evaluate the diagnostic performance of the test TRAP-myelin
Sponsor: Nantes University Hospital (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BRD/10/06-S; 2010-A00892-37 (Other: ANSM)
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2014-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; TRAP; TRAP-Myéline
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Relapsing Multiple Sclerosis- group 1 (Other): Definite multiple sclerosis according to the McDonald criteria, relapsing Patient innocent of thorough treatment or treatment immunomodulator stopped for at least 6 months.
  Interventions: Device: Trap Myelin Test
- Relapsing Multiple Sclerosis- group 2 (Other): Multiple sclerosis defined according to the criteria of McDonald, relapsing Patient under treatment immunomodulator for at least 6 months.
  Interventions: Device: Trap Myelin Test
- secondary progressive multiple sclerosis- Group 3 (Other): Multiple sclerosis defined according to the criteria of McDonald, secondary progressive multiple sclerosis
  Interventions: Device: Trap Myelin Test
- primary progressive multiple sclerosis- group 4 (Other): Multiple sclerosis defined according to the criteria of McDonald, primary progressive multiple sclerosis
  Interventions: Device: Trap Myelin Test
- control 1 (Other): healthy volunteers
  Interventions: Device: Trap Myelin Test
- Control 2 (Other): Patients with central or peripheral neurological non-inflammatory, non-autoimmune.
  Interventions: Device: Trap Myelin Test
- Control 3 (Other): Patients having an autoimmune pathology
  Interventions: Device: Trap Myelin Test

INTERVENTIONS:
Device: Trap Myelin Test

SUMMARY:
The objective of this project is to characterize the response TRAP positive patients with Multiple Sclerosis (MS) and to evaluate the sensitivity and specificity of the method in order to develop a second time as a diagnostic tool in this disease. We plan to analyze the response TRAP over a hundred patients with various clinical stages SEP (relapsing, progressive forms) and compared to healthy controls,

ELIGIBILITY:
Inclusion Criteria:

* These criteria depend on the subgroup belongs to the patient.
* Signed consent
* Membership of a social security system

Exclusion Criteria:

* Whatever the patient group or control:
* Processing immunosuppressive.
* Processing by a monoclonal antibody.
* Previous treatment with an immunosuppressant for a significant period of time (more than 6 months of oral treatment, more than 6 cycles of cyclophosphamide over 3 cures mitoxantrone).
* Carcinomatous pathology known evolving.
* People under guardianship.
* Pregnant women.
* Patients not motivated to study. Known patients with anemia (hemoglobin <10g/100ml)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 189 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the diagnostic performance of myelin-TRAP assay for Multiple Sclerosis | 2 years
  The main criterion corresponds to the area under the curve ROC (Receiver operating characteristic). The curve ROC is a graphic representation of the existing relation between the sensibility and the specificity of a test, calculated for all the values possible thresholds. The performance of the test TRAP-myéline will thus be estimated by means of the area calculated under this curve

SECONDARY OUTCOMES:
Determine the best cut-off rate of myelin-Trap and evaluate the sensitivity and specificity associated | 2 years

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - University Hospital of Bordeaux, Bordeaux
  - Hopital neurologigue Pierre Wertheimer, Bron
  - University Hospital of clermont Ferrand, Clermont-Ferrand
  - University Hospital of Lille, Lille
  - University Hospital of Marseille, Marseille
  - University Hospital of Montpellier, Montpellier
  - University Hospital of Nantes, Nantes
  - University Hospital of Nice, Nice
  - University Hospital of Rennes, Rennes
  - University Hospital of Strasbourg, Strasbourg
  - University Hospital of Toulouse, Toulouse